CLINICAL TRIAL: NCT00417742
Title: A Randomized Trial of Headache Management Programs
Brief Title: Project CHEER (Comprehensive Headache Evaluation, Education, Relief)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Innovative Medical (Industry); Thomas Jefferson University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0728; AHRQ Grant No.: 1 R01 HS10893; 0728-06-5R7ER
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Headache
Keywords: headache; migraine headache; tension headache
MeSH Terms: conditions — Headache Disorders; Headache; Migraine Disorders; Tension-Type Headache

INTERVENTIONS:
Behavioral: Service delivery through a Headache Management Program

SUMMARY:
PROJECT CHEER is a randomized controlled trial designed to test the effectiveness of a comprehensive focused approach to headache care. Three institutions are collaborating in this trial by establishing special Headache Programs that can provide individualized treatment and follow-up: Duke University Medical Center in Durham, NC; Thomas Jefferson University in Philadelphia, PA; and Kaiser Permanente in San Diego, CA. Support and oversight are provided by the U.S. Agency for Healthcare Research and Quality.

HEADACHE sufferers age 18 and over whose headaches interfere with their ability to work, study or enjoy life are eligible for this trial. Half of the enrolled individuals will be selected at random to receive care in the Headache Program and half will continue to receive care as usual from their primary care providers.

EVALUATION is an important part of this project. Every participant completes a screening interview and survey at the time of enrollment. The initial evaluation will provide an accurate diagnosis of headache type(s). The results of this evaluation will be reported to the primary care provider and may help to provide usual care. Subjects assigned to the Headache Program are further evaluated by the program manager in consultation with a headache specialist.

EDUCATION in headache care is provided to participants assigned to the Headache Program.

The classes include suggestions on diet and lifestyle as well as a review of medication use.

Note: The above is excerpted from the flyer we distributed to recruit patients to the trial.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether headache management programs should be promoted as a preferred strategy for managing patients with chronic disabling headache.

Chronic headache affects between 6% and 17% of the population and is associated with significant numbers of days lost from work and reduced quality of life, as well as disproportionate use of medical resources. Current treatment is sub-optimal, with patients often not adequately diagnosed and/or not receiving appropriate preventive and acute pharmacologic therapy or behavioral modification. As a result, chronic headache is associated with sub-optimal quality of care, high patient dissatisfaction as well as high cost to individuals, insurers, and society.

The specific hypothesis of this study is that a properly designed headache management program (HMP) will reduce headache-related disability, improve process of care, and reduce management costs for patients with chronic headache. The format is a randomized controlled trial in which a patient population participating in a HMP will be compared with a corresponding patient population receiving usual care. A pilot study1 has determined the components of an optimal HMP and the effectiveness of a prototype of this service with a limited number of patients at a Kaiser Permanente facility in Santa Rosa, California.

ELIGIBILITY:
Inclusion Criteria:

* age 21 or over
* have chronic headache thought to be of tension-type, migraine or mixed etiology
* intend to continue headache care at their current location for the next six months
* MIDAS score >5

Exclusion Criteria:

* Under age 21
* Currently seeing a neurologist for headache care
* Currently being seen in a Headache Clinic
* MIDAS score <5

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828
Dates: Start 2002-06; Study Completion 2004-12

PRIMARY OUTCOMES:
MIDAS, simple and accurate five-question survey that measures days lost to headache disability during the last 3 months and also headache pain on a 10-point scale.
The measure is taken by telephone at the screening interview and by mailed survey at basel

SECONDARY OUTCOMES:
CATI headache diagnostic survey is administered by telephone at the screening interview to obtain a diagnosis of headache type.
SF-36 Quality of Life Survey is administered by mailed survey at baseline and at 6 and 12 months
Health Care Utilization Measures will include self-report by patients on the mailed surveys at baseline and at 3, 6 and 12 months.
Patients are asked about their use of outpatient, inpatient and emergency room services, as well as use of alternative therapies (e.g., accupuncture, massage therpay, herbalists) and prescription and nonprescription drugs.
Patient reports will be validated by administrative utilization data and by a limited chart review at each site.

CONTACTS AND LOCATIONS:
Overall Officials: David B Matchar, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Kaiser Permanente, San Diego, California
  - Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Harpole LH, Samsa GP, Jurgelski AE, Shipley JL, Bernstein A, Matchar DB. Headache management program improves outcome for chronic headache. Headache. 2003 Jul-Aug;43(7):715-24. doi: 10.1046/j.1526-4610.2003.03128.x. PMID 12890125